CLINICAL TRIAL: NCT05420571
Title: Application of Digital Impression Technology in Children's Dental Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022（59）
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Dental Trauma
Keywords: Immature permanent teeth ；Dental Trauma；Digital impressions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital impression module (Experimental): In the experimental group, digital impressions and 3D printed models were used and fitted pads were made. Patients were instructed to wear the hinge pad for 24 hours, and x-rays were taken and intraoral examinations were performed at 2 weeks and 4 weeks.
  Interventions: Procedure: digital impression
- ordinary impression group (Active Comparator): The control group used alginate impression and plaster model infusion to make the model and make the fitting pad. Patients were instructed to wear the pad for 24 hours, and x-rays and intraoral examinations were taken at 2 and 4 weeks.
  Interventions: Procedure: alginate impression

INTERVENTIONS:
Procedure: digital impression — 3D printed models after digital impressions
  Arms: digital impression module
Procedure: alginate impression — Alginate impressions after plaster model infusion to make models
  Arms: ordinary impression group

SUMMARY:
We will Choose patients with tooth loosening caused by tooth trauma and requiring fix in the department of Pediatric Dentistry and emergency of Stomatology Hospital, Zhejiang University School of Medicine, from July 2022 to May 2025. These patients will be randomly divided into digital impression module (experimental group) and ordinary impression group (control group).The operation time, comfort index and efficacy index of the two groups were compared to investigate the advantages of digital impressions in the application of traumatic dental injuries in children.

DETAILED DESCRIPTION:
1. Information on medical history, physical examination, and ancillary tests were collected and recorded by the pediatric dentistry and emergency department to determine the inclusion subjects, and the grouping was determined according to a randomized controlled design.
2. In the experimental group, digital impressions + 3D printed models were used and fitted pads were made; in the control group, alginate impressions + plaster model infusion were used to make models and fitted pads were made. The included subjects were routinely examined intraorally before and after treatment. Patients were instructed to wear the hinge pad for 24 hours and X-ray films were taken and intraoral examination was performed at 2 weeks and 4 weeks.
3. The observation indexes included： (1) operation time: operation time for the child's chair position, (2) comfort index: pain assessment of patients using visual analog scale, (3) efficacy indexes: a. tooth sensitivity, gingival margin irritation, and lip irritation were assessed using visual analog scale (VSA); B. fixation efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years old ② Loosening or dislocation of anterior teeth caused by trauma; ③ Degree I, II and III of tooth mobility, excluding normal physiological mobility; ④ No jaw fracture, root fracture, avulsion injury and individual malocclusion; ⑤ Children can cooperate with treatment and follow up on time

Exclusion Criteria:

① Children have clear systemic disease factors (various syndromes, hormone level disorders, metabolic diseases, etc.); ② Patients with periodontal disease; ③ Children or family members do not agree to participate in the study; ④ Uncooperative or intolerable examination and treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Fixed efficiency | four weeks
  Fixed effective as the affected tooth loosening does not exceed the physiological degree of movement, X-ray examination periodontal membrane without widening without abnormal shadow of the root tip

CONTACTS AND LOCATIONS:
Overall Officials: LinXian Fang, Master, Principal Investigator — The Stomatology Hospital, Zhejiang University School of Medicine
Locations (1):
- The Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China